CLINICAL TRIAL: NCT00019864
Title: Osteosarcoma: Outcome of Therapy Based on Histologic Response. A Collaborative Effort of the POB/NCI, Texas Children's Hospital and University of Oklahoma.
Brief Title: Combination Chemotherapy Before and After Surgery in Treating Patients With Osteosarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067263; NCI-99-C-0125I; NCT00001821 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2007-10

CONDITIONS: Cardiac Toxicity; Sarcoma
Keywords: cardiac toxicity; localized osteosarcoma; metastatic osteosarcoma; recurrent osteosarcoma
MeSH Terms: conditions — Cardiotoxicity; Sarcoma; Osteosarcoma | interventions — Filgrastim; Cisplatin; Dexrazoxane; Doxorubicin; Leucovorin; Methotrexate; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: dexrazoxane hydrochloride
Drug: doxorubicin hydrochloride
Drug: leucovorin calcium
Drug: methotrexate
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy before surgery may shrink the tumor so that it can be removed during surgery. Giving chemotherapy after surgery may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving chemotherapy before and after surgery works in treating patients with osteosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the rate of in vivo histologic response in patients with osteosarcoma treated with neoadjuvant cisplatin, methotrexate, and doxorubicin with dexrazoxane (as cardioprotection).
* Determine the event-free and overall survival of patients with nonmetastatic disease who show good response to neoadjuvant therapy and receive adjuvant therapy with the same regimen.
* Determine the event-free survival of patients with nonmetastatic disease who show poor response to neoadjuvant therapy and receive adjuvant therapy with the same regimen.
* Determine the event-free survival and overall survival of patients with metastatic disease who receive neoadjuvant therapy.

OUTLINE: This is a multicenter study.

* Neoadjuvant therapy: Patients receive neoadjuvant chemotherapy comprising dexrazoxane IV over 15 minutes, doxorubicin IV over 15 minutes, and cisplatin IV over 4 hours on days 1 and 2 in week 0. Patients also receive methotrexate IV over 4 hours followed by leucovorin calcium in weeks 3 and 4. Patients then receive filgrastim (G-CSF) subcutaneously (SC) once daily beginning 24 hours after completion of chemotherapy and continuing until blood counts recover. Treatment repeats every 5 weeks for 2 courses in the absence of disease progression or unacceptable toxicity.
* Surgical resection: Patients undergo definitive surgery in week 11.
* Adjuvant therapy: Patients receive dexrazoxane, doxorubicin, cisplatin, methotrexate, and leucovorin calcium as in neoadjuvant therapy*. Treatment repeats every 5 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *Cisplatin is not administered in courses 3 and 4 of adjuvant therapy

Patients are followed within 4 weeks, every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed osteosarcoma

  * No more than 1 month since prior diagnostic biopsy
  * Nonmetastatic malignant high-grade osteosarcoma of bone
  * Histologically confirmed metastatic disease allowed
  * Unresectable primary disease allowed
* No low-grade, parosteal, or periosteal osteosarcoma

PATIENT CHARACTERISTICS:

Age:

* 25 and under

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8.0 g/dL

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* ALT less than 5 times normal

Renal:

* Creatinine no greater than 1.5 times normal
* Creatinine clearance or radioisotope glomerular filtration rate greater than 70 mL/min

Cardiovascular:

* Shortening fraction at least 27% by echocardiogram or MUGA
* Ejection fraction at least 45% by echocardiogram or MUGA

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* Not specified

Other:

* No other concurrent therapy with no evidence of progressive disease

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2000-03; Primary Completion 2006-12 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Rate of in vivo histologic response
Event-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi Dagher, MD, Study Chair — National Cancer Institute (NCI)
Locations (4):
- United States (4):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas